CLINICAL TRIAL: NCT03018795
Title: The Effect of Ozone Therapy as an Adjunct to the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial
Brief Title: Ozone Therapy as an Adjunct to the Surgical Treatment of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25901600-2858
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; Surgical regenerative treatment; ozone therapy
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ozone Group (Active Comparator): Decontamination of implant surfaces with saline irrigation and additional ozone therapy in combination with regenerative surgery
  Interventions: Procedure: Decontamination of implant surfaces
- Control Group (Active Comparator): Decontamination of implant surfaces with saline irrigation alone in combination with regenerative surgery
  Interventions: Procedure: Decontamination of implant surfaces

INTERVENTIONS:
Procedure: Decontamination of implant surfaces — Decontamination of implant surfaces in combination with regenerative surgery

SUMMARY:
Decontamination procedure is a challenging factor that affects the success of surgical regenerative therapy (SRT) of peri-implantitis. The purpose of the present study was to determine the impact of additional ozone therapy for the decontamination of implant surfaces in SRT of peri-implantitis. A total of 21 patients with moderate or advanced peri-implantitis were randomly allocated to the test group (ozone group) with the use of sterile saline with additional ozone therapy or the control group with sterile saline alone for decontamination of the implant surfaces in SRT of peri-implantitis. Clinical and radiographic outcomes were evaluated at baseline and 6 months postoperatively

DETAILED DESCRIPTION:
Peri-implant diseases are described as inflammatory processes in the tissues surrounding implants in response to mainly microbial biofilms on the surface of the implants (Zitzmann and Berglundh 2008). Peri-implant mucositis is described as an inflammatory reaction triggered by microbial biofilms without any loss of peri-implant bone, while peri-implantitis is characterized by bleeding when probed and/or suppuration with further loss of the peri-implant bone (Lindhe and Meyle 2008; Lang and Berglundh 2011).

Since microbial biofilms play a major role in the etiology (Becker et al. 1990; Quirynen et al. 2002), it has been considered that elimination of microbial pathogens is mandatory in the treatment of peri-implant diseases (Mombelli and Lang 1994; Schwarz et al. 2006). The objectives of peri-implantitis therapy are implant surface decontamination to resolve inflammation resolution while preserving the implant supporting tissues (Lindhe and Meyle 2008; Heitz-Mayfield and Lang 2010).

Several implant decontamination methods have been suggested, including mechanical debridement, chemical therapy (applications of root conditioners, disinfectants, and local and systemic antibiotic therapy) (Heitz-Mayfield et al. 2012; Wohlfahrt et al. 2012) and surgical procedures aiming to remove bacteria, and smooth, decontaminate and detoxify the implant surface (Froum et al. 2012; Schwarz et al. 2013). However, there is as yet no consensus on the most effective protocol for implant surface detoxification (Suarez et al. 2013).

Ozone has a strong oxidation effect with remarkable antimicrobial potential and can be used as a disinfectant in clinical applications of dentistry (Iliadis and Millar 2013). A previous study reported that ozone has powerful antimicrobial activity in response to anaerobic periodontal pathogenic microorganisms and may have the potential to be used as an adjunctive tool in non-surgical periodontal therapy in periodontitis patients (Eick et al. 2012). Ozone therapy can promote haemostasis, enhance the release of growth factors and local oxygen supply, upregulate cellular antioxidant enzymes and inhibit bacterial proliferation (Ozdemir et al. 2013). However, current literature has little information regarding the antimicrobial activity of ozone in the treatment of peri-implant diseases. A previous randomized, clinical study showed that ozone therapy reduced inflammation in the treatment of peri-implant mucositis (McKenna et al. 2013). Another in-vitro trial reported that in the reduction of adherent bacteria on titanium, gaseous ozone showed selective efficacy without any adverse effect on the surface structures of the titanium surfaces or the adhesion and proliferation of osteoblastic cells (Huser-Gerspach et al. 2012).

Non-surgical therapy alone has been reported to be inadequate for the treatment of moderate and severe forms of peri-implantitis and therefore surgical therapy is frequently required (Lindhe and Meyle 2008). The goals of surgical therapy of peri-implantitis are mainly to be able to access areas for mechanical debridement and implant surface decontamination and to reconstruct the anatomic conditions to improve plaque control and to eliminate the pathological peri-implant pockets (Esposito et al. 2012; Roos-Jansaker et al. 2014). This can be achieved with resection or with procedures of bone regeneration such as guided bone regeneration (Roos-Jansaker et al. 2003; Schou et al 2004; Sahrmann et al. 2011).

Studies have evaluated the combination of various regenerative biological agents and techniques for surgical regenerative therapy (SRT) of peri-implantitis and clinical and radiological improvements following different bone augmentation procedures have been reported (Claffey et al. 2008; Schwarz et al. 2009; Roos-Jansaker et al. 2011; Renvert et al. 2012). A long-term, clinical study demonstrated that vertical peri-implant bone defects (PBDs) may be actively treated by regenerative surgical means, using a bone substitute alone or in combination with a membrane (Roos-Jansaker et al. 2014).

Platelet concentrates are preferred in periodontal surgical procedures for the purpose of accelerating angiogenesis, stimulating the activity of osteoblasts and fibroblasts, and obtaining regeneration of hard and soft tissues, including stem cells and growth factors (Del Fabbro et al. 2011). These materials can be used alone or in combination with bone grafts or barrier membranes. In studies employing bone grafts with the use of platelet rich fibrin (PRF) or PRF alone around PBDs it has been reported that PRF leads to increased new bone formation and a higher bone to implant contact ratio (Lee et al. 2012; Simsek et al. 2016). A recent study reported that treatment of peri-implantitis using PRF was clinically more effective than with access flap surgery alone. It was also concluded in the study that PRF improves the outcomes of surgical peri-implantitis treatment (Hamzacebi et al. 2015).

There have been recent developments of various techniques using platelet concentrate to provide different rates of platelets, leukocytes, growth factors, stem cells and fibrin matrix. Sacco developed concentrated growth factors (CGF) as a therapeutic protocol obtained by separating the venous blood centrifuged using a special device in the same manner as PRF (Rodella et al. 2011). It was also argued that centrifugation at a different speed provides a larger, denser fibrin matrix compared to PRF, which results in improved regenerative capacity and greater versatility (Sohn et al. 2009). Some recent studies have reported that CGF accelerates new bone formation related to guided bone regeneration (Sohn et al. 2011; Kim et al. 2014).

The purpose of this randomized, controlled clinical study was to evaluate the clinical and radiological results of implant surface decontamination using sterile saline alone or in combination with ozone therapy applied as surgical regenerative treatment for peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years,
2. presence of peri-implantitis exhibiting one of the defect configurations as defined by either a Class Ib (buccal dehiscence + semicircumferential bone resorption), Class Ic (i.e. buccal dehiscence + circular bone resorption) or Class Ie (i.e. circumferential bone resorption) with a probing depth of >6 mm
3. radiographic bone loss ≥2 mm on at least at one implant surface,
4. peri-implant sites with bleeding or suppuration after probing,
5. no implant mobility,
6. no evidence of occlusal overload
7. non-smoker.

Exclusion Criteria:

1. serious systemic disease that would contraindicate for periodontal surgery (i.e. diabetes (HbA1c < 7),
2. prophylactic antibiotics required or systemic antibiotic administration during the past 3 months, and (3) placement, and prosthetic loading of implants within the past 1 year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
probing depth of peri-implantitis sites | 6 months postoperatively
  measured as the distance between the deepest site of the pocket to the peri-implant mucosal margin

SECONDARY OUTCOMES:
bone loss of peri-implant defects | 6 months postoperatively
  Measurements were taken of mesial and distal distances between the first bone to implant contact and bone loss (BL) in the implant shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Berrin Unsal, PhD, Study Director — Prof Dr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isler SC, Unsal B, Soysal F, Ozcan G, Peker E, Karaca IR. The effects of ozone therapy as an adjunct to the surgical treatment of peri-implantitis. J Periodontal Implant Sci. 2018 Jun 30;48(3):136-151. doi: 10.5051/jpis.2018.48.3.136. eCollection 2018 Jun. PMID 29984044